CLINICAL TRIAL: NCT04460235
Title: Immunogénicité de la Vaccination Anti-pneumococcique (PCV13+PPV23 Versus PREVENAR20) Dans le Lymphome Chez l'Adulte
Brief Title: Clinical Trial Assessing the Immunogenicity of an Anti-pneumococcal Vaccination Strategy (PCV13+PPV23 Versus PREVENAR20) in Adult Patients Treated for a Lymphoma
Acronym: HEMATOVAC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HEMATOVAC; 2024-517288-22-01 (EU CTIS Number)
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Vaccine; Streptococcus Pneumoniae; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — 13-valent pneumococcal vaccine; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort study A (Other): 80 patients already included in study cohort A. They received an injection of 13-valent conjugate vaccine (PCV13), followed by an injection of 23-valent polysaccharide vaccine (PPV23) at least 2 months later.
  Interventions: Biological: Prevenar 13 + Pneumovax 23
- Cohort study B (Other): 80 patients to be included in study cohort B. They will receive a single injection of PREVENAR20 vaccine.
  Interventions: Biological: PREVENAR20

INTERVENTIONS:
Biological: Prevenar 13 + Pneumovax 23 — Cohort study A before modification of vaccination national guidelines
  Arms: Cohort study A
Biological: PREVENAR20 — Health authorities changed guidelines to recommend one injection of PREVENAR20 instead of the 2-vaccine scheme general practitioners are usually in charge of this vaccination.
  Cohort study B
  Arms: Cohort study B

SUMMARY:
The French Public Health Council recommended pneumococcal vaccination combined strategy for all immunocompromised patients in 2012. This strategy consisted in conjugated 13-valent pneumococcal (PCV13) injection followed 2 months later by polysaccharide 23-valent (PPV23) vaccine injection. In 2024, Health authorities changed guidelines to recommend one injection of PREVENAR20 instead of the 2-vaccine scheme general practitioners are usually in charge of this vaccination. Conjugated pneumococcal vaccine enhances the immunogenicity of the polysaccharide vaccine. Acute leukemia and lymphoma are treated with multiple courses of chemotherapy, impairing the immune system and potentially the response to vaccination. These patients are more at risk for developing pneumococcal invasive diseases than the general population. However, efficacy of pneumococcal vaccination is poorly documented in this setting. We assume that 65% of the patients are non-responders to double compared to 45% for PCV20PREVENAR20 vaccination, according to their anti-pneumococcal immunoglobulin G (Ig) titers and the opsonophagocytic activity (OPA). To assess the immunogenicity of the pneumococcal vaccination combined strategy in adult population of acute leukemia and lymphoma, we will measure anti-pneumococcal serotype-specific IgG titers and OPA at different time-points after completion of the combined vaccine strategy. The primary objective is to assess the immunogenicity of pneumococcal vaccination combined strategy at 3 months after the PCV13 injection (corresponding to 1 month after the end of the combined strategy in cohort A) using Ig G titers and OPA, compared to 3 months post PREVENAR20 (cohort B). At different time points (day 0, 4 weeks post PCV13, and 4 weeks, 3-6 months and 9-12 months post PPV23 and in day 0, 4 weeks post PREVENAR20 and 3 months, 5-8 months and 11-14 months post PREVENAR20, the immunological response to vaccination will be monitored using specific-serotype IgG titers, OPA, and total anti-pneumococcal Ig. We will determine predictive factors of non-response to vaccination by comparing demographic data, biological data and treatment received lymphoma patients. The tolerance and safety of the vaccination strategy will also be assessed in this specific hematological population.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 year-old.
* AND medical follow-up in hematology unit
* AND had received a first course of chemotherapy for diffuse large B cell lymphoma or for follicular lymphoma
* Life expectancy > 6 months.
* Negative pregnancy test.
* Having signed the consent form.
* Having an health insurance.

Exclusion Criteria:

* Receiving monoclonal antibodies or biotherapies altering the immune response, other than anti-CD20 antibodies in the chemotherapy protocol.
* Uncontrolled bacterial, viral or fungal infection less than 7 days.
* Previous vaccination with PCV13 or PPV23 (unless PCV13 was administered in childhood. The last injection must be performed at least five years ago).
* Preexisting condition that altered the immune response: splenectomy, HIV, primary or secondary immune deficiency, nephrotic syndrome, sickle cell anemia, autoimmune disorder, solid organ transplantation, immunosuppressive drugs or biotherapy not included in the chemotherapy.
* Patient who already received chemotherapy for malignancy in the previous 2 years before the inclusion.
* Major blood clotting disorders preventing intramuscular injection.
* Medical history of anaphylactic reaction to vaccination.
* Known allergy to one of the vaccine components.
* Involvement to another vaccine biomedical research.
* Protected person.
* Pregnant women or women of childbearing age without appropriate contraceptive measures.
* Perfusion of polyvalent immunoglobulins during follow-up.
* Participants with hypersensitivity to aluminum phosphate, phenol or CRM197 protein, protein derived from Corynebacterium diphtheria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients having an immunological response | 4 weeks after the end of the combined strategy for cohort study A and 3 months post injection for cohort study B
  Proportion of patients having an immunological response to combined strategy at 4 weeks after the end of the combined strategy compared to proportion of patients having an immunologicalresponse at 3 months post PREVENAR20 injection.
  An immunological response to vaccination is defined by 7/10 tested serotypes responding to these 4 criteria: a serotype-specific IgG titer ≥ 1,3 μg/mL (WHO threshold), a two-fold increase of this IgG titer compare to baseline before vaccination, a serotype-specific OPA ≥1/8, and a four-fold increase of functional antibodies compare to baseline.

SECONDARY OUTCOMES:
Proportion of patients having an ELISA serotype-specific IgG titer and a two-fold increase of this IgG titer | 4 weeks after injection
  Proportion of patients having an ELISA serotype-specific IgG titer ≥ 1.3 μg/mL (WHO threshold) and a two-fold increase of this IgG titer compared to baseline at 4 weeks after the PCV13 or PREVENAR20 injection
Proportion of patients having a sustainable response to vaccination | 3-6 months after the PPV23 injection or 5-8 months post PREVENAR20
  Proportion of patients having a sustainable response to vaccination defined by an ELISA serotype-specific IgG titer ≥ 1μg/mL (WHO threshold) and a two-fold increase of this IgG titer compared to baseline between 3-6 months after the PPV23 injection or 5-8 months post PREVENAR20.
Proportion of patients having a sustainable response to vaccination | 9-12 months after the PPV23 injection or 11-14 months post PREVENAR20.
  Proportion of patients having a sustainable response to vaccination defined by the same criteria as the primary outcome and measured between 9-12 months after the PPV23 injection or 11-14 months post PREVENAR20.
Proportion of responding patients having titers of IgG, IgG2, IgM, and IgA rising significantly | 4 weeks after PCV13 or PREVENAR20 injection, and 4 weeks, 3-6 months and 9-12 months after PPV23 injection versus respectively 3 months, 5-8 months and 11-14 months after PREVENAR20 injection.
  Proportion of responding patients having titers of IgG, IgG2, IgM, and IgA rising significantly at 4 weeks after PCV13 or PREVENAR20 injection, and 4 weeks, 3-6 months and 9-12 months after PPV23 injection versus respectively 3 months, 5-8 months and 11-14 months after PREVENAR20 injection.
  A significant increase is defined by a 4-fold increase of IgG and IgG2 titers, a 13-fold increase of IgA titers, and a 20-fold increase of IgM titers compared to baseline at inclusion.
Predictive factors for non-response to vaccination | 4 weeks, and 9-12 months after PPV23 versus respectively 3 months and 11-14 months after PREVENAR20 injection
  To determine predictive factors for non-response to vaccination at 4 weeks, and 9-12 months after PPV23 versus respectively 3 months and 11-14 months after PREVENAR20 injection such as age, immune status, chemotherapy, immunotherapy.
Local or general reactions to vaccination and invasive pneumococcal infections | 14 months
  Number of patients having local or general reactions to vaccination and number of invasive pneumococcal infections with a documented serotype considered as vaccination failure.
Concordance between the reference immuno-monitoring dosage and another kit of dosage | 14 months
  To assess the concordance between the reference immuno-monitoring dosage (WHO ELISA) and another kit of dosage (Vacczyme® Binding Site®).

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Chu Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU Limoges, Limoges
  - Chu Nantes, Nantes
  - Ch Perigueux, Périgueux
  - CHU Poitiers, Poitiers
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided
Undecided